CLINICAL TRIAL: NCT05257564
Title: Performance and Usability Evaluation of Cardiometabolic Point-of-care Devices in a Target Use Setting
Brief Title: Cardiometabolic Devices Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University Hospital, Geneva (Other); B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NC001
Record Dates: First submitted 2022-01-28; First posted 2022-02-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases; Hyperlipidemias
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Prospective quantitative accuracy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Other): Fingerstick collection and venous whole blood collection.
  Interventions: Device: Determine the accuracy of quantitative measurements of GLU, HbA1c,CHOL and CRE with POC devices compared to a laboratory reference method (Roche)

INTERVENTIONS:
Device: Determine the accuracy of quantitative measurements of GLU, HbA1c,CHOL and CRE with POC devices compared to a laboratory reference method (Roche) — Fingerstick capillary blood will be collected according to each manufacturer's Instructions for use. The fingerstick capillary blood samples will be used immediately on the point-of-care assays. The venous blood will be collected in specific tubes for plasma (GLU), for whole blood (HbA1c) and for serum (CREP, CHOL). Plasma will be separated by centrifugation at the PHC facility and health post and aliquots will be prepared. Serum will be left to clot prior to centrifugation and serum aliquots will be prepared at the PHC facility and health post. The samples will be stored until transfer to the BPKIHS reference lab.

SUMMARY:
With the rise of cardiovascular diseases (CVD) and diabetes, the global disease burden is shifting towards non-communicable diseases (NCDs). An increasing number of low- and middle-income countries (LMICs) are currently experiencing the double burden of infectious and non-communicable diseases. In order to facilitate a patient-centred approach to healthcare, there is an urgent need to ensure that primary healthcare (PHC) facilities in LMICs are capable of addressing diagnosis and monitoring of non-communicable diseases at the point-of-care (POC). Important minimum parameters for PHC POC diagnosis and monitoring of cardiometabolic diseases are lipids/lipoproteins, glucose, glycated haemoglobin (HbA1c) and serum creatinine, to address cardiovascular disease, diabetes and chronic kidney disease.

While several technologies of multi-parameter POC devices capable of supporting diagnosis and monitoring of cardiometabolic diseases exist, their quantitative accuracy is often not well evaluated outside of the manufacturer's laboratories and published independent evaluations can be rare, particularly in the settings of intended use. These settings are PHC facilities in varying climatic environments and with staff without specialist laboratory training. Our study aims to evaluate the quantitative accuracy of 2 cardiometabolic POC devices in a setting of intended use and performed by the intended user. (Evaluating the quantitative measurements of glucose, HbA1c, total cholesterol and creatinine as measured in a healthcare setting with point-of-care multiparameter devices compared to a laboratory reference method).

DETAILED DESCRIPTION:
Independent performance evaluation of POC devices have shown that many devices, regardless of their intended use, do not perform as well as the manufacturers' claims may suggest. There are a variety of reasons for this, including difference in skills levels of personnel who were involved in generating the data for the manufacturer's claims and who actually perform the test in a clinic, limited evaluation of samples from different geographical locations and thus potential interfering substances or less controlled environmental conditions (e.g. dust, heat and humidity).

Independent performance evaluations to assess clinical accuracy, as well as system usability are important to drive adoption of any technology, and even more so, if the technology is intended to move testing outside of the traditional setting, i.e. away from the central laboratory to the point-of-care. Many devices appear ideally suited for certain settings, however when it comes to actual implementation, the users often discover that the device and workflow do not meet their needs. The choice of a suboptimal device means badly invested resources and may lead to inappropriate use, resulting in fewer reliable tests for patients in the absence of alternatives. Data from real-world evaluations in settings of the intended use can support decision makers to select the right device.

The setting for this study will be a primary healthcare facility and a health post in Nepal, where study participants attend the facility in the context of the "Early detection and management of Chronic Kidney Diseases, Hypertension, Diabetes and Cardiovascular disease in Community in Nepal (KHDC-Nepal) program", conducted by the University Hospital of Geneva and the BP Koirala Institute of Health Science in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older (in line with KHDC eligibility age)
* Attending the Dhulabari PHC facility or Kakarvitta health post in the context of the KHDC program
* Haemoglobin levels ≥8 g/dL
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to provide sufficient capillary or venous whole blood sample for all tests
* Haemoglobin levels < 8g/dL
* Anyone attending the Dhulabari PHC facility or Kakarvitta health post for other reasons than the KHDC program

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation estimation of quantitative measurements of cardiometabolic blood parameters measured on a point-of-care device versus a laboratory reference method | 4 months
  Estimates of correlation between quantitative measurements of blood glucose, HbA1c, total cholesterol and creatinine collected from capillary blood and tested with point-of-care multiparameter devices versus quantitative measurements of blood glucose, HbA1c, total cholesterol and creatinine collected from venous blood and tested with a laboratory reference method.
Limits of agreements estimation of quantitative measurements of cardiometabolic blood parameters measured on a point-of-care device versus a laboratory reference method | 4 months
  Estimates of limits of agreement for quantitative measurements of blood glucose, HbA1c, total cholesterol and creatinine collected from capillary blood and tested with point-of-care multiparameter devices versus quantitative measurements of blood glucose, HbA1c, total cholesterol and creatinine collected from venous blood and tested with a laboratory reference method.

SECONDARY OUTCOMES:
Operational characteristics of study device Tascom | 4 months
  Rate of invalid test results and error types for Tascom (POC device)
Operational characteristics of study device JanaCare | 4 months
  Rate of invalid test results and error types for JanaCare(POC device)
Usability of study devices Tascom | 4 months
  System usability score for Tascom (POC device) SUS Score (>80.3, Grade A, Excellent) SUS Score (68-80.3, Grade B, Good) SUS Score (68, Grade C, Okay) SUS Score (51-68, Grade D, Poor) SUS Score (<51, Grade F, Awful)
Usability of study devices JanaCare | 4 months
  System usability score for JanaCare(POC device) SUS Score (>80.3, Grade A, Excellent) SUS Score (68-80.3, Grade B, Good) SUS Score (68, Grade C, Okay) SUS Score (51-68, Grade D, Poor) SUS Score (<51, Grade F, Awful)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Sharma, Prof.Dr, Principal Investigator — head of the B.P Koirala Institute of Health Sciences
Locations (1):
- B.P Koirala Institute of Health Sciences, Dharān, Sunsari, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giachino M, Vetter B, Perone SA, Correia JC, Erkosar B, Heller O, Khanal VK, Lab B, Pataky Z, Poudel S, Rai M, Sharma SK. Performance and usability of cardiometabolic point of care devices in Nepal: A prospective, quantitative, accuracy study. PLOS Glob Public Health. 2024 Oct 3;4(10):e0003760. doi: 10.1371/journal.pgph.0003760. eCollection 2024. PMID 39361597

DOCUMENTS (1):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT05257564/Prot_000.pdf